CLINICAL TRIAL: NCT07105189
Title: Feasibility of Wireless Continuous Vital Sign Monitoring and Impact on Patients Undergoing Adult Spinal Surgery in a General Ward
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Camilla Hedegaard Larsen, Clinical nurse specialist and Ph.d-student, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: WCVSM-ASD
Record Dates: First submitted 2025-01-10; First posted 2025-08-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Adult Spinal Deformity; Wireless Continuous Vital Signs Monitoring; Wireless Vital Signs Monitoring System; Acceptability; ASD Surgery; Remote Monitoring; Feasibility Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wireless continuous vital sign monitoring in patients undergoing adult spinal deformity surgery (Experimental): Participants in this arm will receive a wearable wireless continuous vital sign monitoring system (CPC12S), applied after spinal deformity surgery and worn during the initial postoperative period (typically 3-5 days). The device transmits data wirelessly to a mobile application accessed by nursing staff.
  Interventions: Device: Wireless monitoring

INTERVENTIONS:
Device: Wireless monitoring — Patients included in the study will be continuous monitored by CPC12S is a wearable sensor that is worn on the chest using electrodes measuring electrocardiography single lead (ECG), Heart rate, respiratory rate, SpO2, blood pressure and temperature.
  The system calculates the heart rate by analysing R-peaks of QRS-complexes in the raw ECG data.
  Respiratory rate is recorded using impedance pneumography. SpO2 is determined by analysing the photoplethysmogram (PPG) wave. Blood pressure is derived by calculating the pulse transit time (PTT) using R-peaks from the QRS complexes, peaks in the photoplethysmogram (PPG) pulse waves, and timing of the second heart-tone corresponding to the dicrotic notch, measured by a stethoscope in the device.
  Temperature is measured by a thermistor placed in the axilla. Vital signs are updated every 20 seconds and measurements are transmitted via Bluetooth to an Android cell phone that is uploading the data via WIFI to a secured server.

SUMMARY:
The goal of this feasibility study is to explore the use of wireless continuous vital sign monitoring in an orthopaedic setting among orthopaedic nurses and patients undergoing adult spinal deformity surgery. In addition to the standard care National Early Warning Score the participants in this study will be monitored by CPC12S a wearable sensor that is worn on the chest using electrodes measuring electrocardiography single lead (ECG), Heart rate, respiratory rate, SpO2, blood pressure and temperature.

Main hypotheses:

The use of wireless continuous vital sign monitoring in daily clinical practice for patients undergoing ASD surgery is feasible in terms of increased acceptability among orthopeadic surgical nurses measured over 12 months with a response rate of at least 80% with an average score of ≥5 at the last measurement in each of the four dimensions of the USE questionnaire: Usefulness, ease of use, ease of learning and satisfaction.

The following parameters will be evaluated:

Primary outcome:

1. The feasibility in terms of acceptability of the concept of wCVSM among orthopedic surgical ward nurses.

   Secondary outcomes:
2. The feasibility in terms of acceptability of the concept of wCVSM in patients undergoing ASD surgery.
3. The technical fidelity of wCVSM, assessed by data collected of vital signs, display of alerts to staff nurses and response to the alerts.
4. The frequency of vital sign deviations in patients after ASD surgery using wCVSM compared to NEWS2.
5. Clinical outcomes of patients undergoing ASD surgery including surgical complications, reinterventions, ICU admissions, unplanned ward transfer, and admissions to another department.

DETAILED DESCRIPTION:
Patients undergoing adult spinal deformity surgery (ASD) is associated with high complication rate and long postoperative recovery (Bess et al., 2023). Patients undergoing ASD surgery are particularly susceptible to adverse events such as electrolyte imbalance, cardiac arrhythmia, anemia, hypotension, fever of unknown origin (Karstensen et al., 2016; Solumsmoen et al., 2021). Additionally, patients undergoing ASD surgery is also associated with severe postoperative pain, often requiring high levels of pain medication (Lamperti et al., 2017; Waelkens et al., 2021), there can lead to decreased respiration rate, sedation, and dizziness (Benyamin et al., 2008).Patients undergoing ASD surgery have a readmission percent within 30 days of 11,8 % and a 2-year all-cause mortality of 3% (Bari et al., 2020).

To ensure safety in patients undergoing ASD surgery, nurses must monitor vital signs to assess patients' health condition and act promptly when signs of clinical deterioration become evident. NEWS2 system is used to identify these early signs of clinical deterioration (Smith et al., 2019). The scoring system relies on six simple physiological parameters, including blood pressure, pulse, respiratory rate, peripheral oxygen saturation, temperature, level of consciousness and an associated algorithm (Smith et al., 2019). Since measurements with NEWS2 are intermittent, they often provide a temporary view of the patient's condition, and the system may therefore overlook changes in the patient's condition that occur between measurement (Downey et al., 2017).

Wireless continuous vital sign monitoring (wCVSM) offers an alternative to intermittent measurements. wCVSM systems can be defined as wearable technologies that enable continuous, real-time vital sign monitoring without direct contact between patients and health-care providers. These systems transmit vital sign data to an application on the nurses´ mobile phones, enabling the recognition of clinical deterioration in real time and facilitating a prompt response to patients' needs (Haahr-Raunkjaer et al., 2022; Leenen et al., 2020). To evaluate the feasibility of wCVSM, it is essential to assess its acceptability among orthopaedic surgical nurses and patients undergoing ASD surgery. Their perceptions and willingness to adopt this technology are essential for ensuring its practical integration, consistent use, and long-term sustainability in enhancing clinical outcomes and patient safety.

This study will contribute to our understanding of wCVSM's potential to enhance patient safety, its applicability in clinical practice, and provide necessary considerations when implementing new technological equipment.

In the current study patients undergoing ASD Surgery will, in addition to standard care the National Early Warning Score 2 (NEWS2) be monitored by wireless continuous vital sign monitoring (wCVSM) using the multiparameter ambulatory telemonitoring system CPC12S system and WARD-CSS application postoperatively.

CPC12S is a wearable sensor that is worn on the chest using electrodes measuring electrocardiography single lead (ECG), Heart rate, respiratory rate, SpO2, blood pressure and temperature. The system can also be used to registration of body position and movement, but this will not be used in this study.

Vital signs are updated every 20 seconds and measurements are transmitted via Bluetooth to an Android cell phone that is uploading the data via WIFI to a secured server.

Once every 20 second the vital signs measurements will be transmitted to the CPC12S software system and when to the WARD application displayed on the electronic device Zebra carried by the nurses. The WARD-CSS application is combining innovative technology with evidence-based algorithms and allow earlier and more frequent detection of patient deterioration trough predictive algorithms (https://ward247.com/wp-content/uploads/2024/11/Instructions-for-Use-WARD-CSS-Version-1.3.x-English-US-v6-20241118_185730.pdf.)

The following parameters will be evaluated:

Primary outcome:

1. The feasibility in terms of acceptability of the concept of wCVSM among orthopedic surgical ward nurses.

   Secondary outcomes:
2. The feasibility in terms of acceptability of the concept of wCVSM in patients undergoing ASD surgery.
3. The technical fidelity of wCVSM, assessed by data collected of vital signs, display of alerts to staff nurses and response to the alerts.
4. The frequency of vital sign deviations in patients after ASD surgery using wCVSM compared to NEWS2.
5. Clinical outcomes of patients undergoing ASD surgery including surgical complications, reinterventions, ICU admissions, unplanned ward transfer, and admissions to another department.

Study design This feasibility study is designed as a single-arm prospective clinical cohort.

Nurse acceptability:

Acceptability by nurses will be measured longitudinally. Acceptability by nurses will be measured by the usefulness, satisfaction, and ease of use questionnaire. The questionnaire is translated into Danish guided by internationally accepted guidelines.

All nurses and nurses' assistants employed on the ward (approx. n=50) will receive the (USE) questionnaire by e-mail at T1 baseline, T2 at 6 months, and T3 at 12 months.

Patient acceptability:

Patient acceptability will be measured cross-sectional by the System Usability Scale (SUS) questionnaire (Brooke, 1995). Patients will receive the SUS questionnaire on paper before discharge.

Fidelity:

Fidelity will be measured prospectively and will focus on the functioning of the continuous monitoring system and will be obtained by analysis of the collected data. Outcomes will be total monitoring time, total number of artefacts (if nonvalid measurement is recorded), number of alerts (system and vital sign), and response to alerts will be assessed using the response buttons on the WARD application.

Frequency of deviations in vital signs in patients after ASD surgery using wCVSM compared to NEWS2 will be measured by following:

1. How many deviations are detected per patient per day with wCVSM.
2. How many deviations are detected per patient per day with NEWS2
3. How often does wCVSM detect deviations that do not appear in NEWS2 measurements.

Clinical outcomes include length of stay, surgical complications according to the Clavien Dindo classification, reinterventions, unplanned ward transfer, and unplanned ICU admissions.

Analysis Data analysis will be conducted using descriptive statistics. Continuous data will be calculated for normal distribution by medians and interquartile or means and standard deviations (SD). Every parameter will be checked for normality by the Shapiro-Wilk test and visually by a histogram. The results from the questionnaires will be analyzed and reported as continuous data.

ELIGIBILITY:
Inclusion Criteria:

* Included are adult patients (>=18 years) scheduled for ASD surgery with estimated a >3 day expected post-operative stay. ASD-surgery is defined as a posterior instrumented fusion of at least five spinal levels including instrumentation to the pelvis, caused by a degenerative condition of the spine.
* Registered nurses and nurses' assistants employed at the orthopedic ward during the study period will be included if they have experience working with wCVSM during the study period. The study includes both sexes, variation of level of education and years of work experience. Included nurses and nurses' assistants should be proficient in the Danish language.

Exclusion Criteria:

* Exclusion criteria are patients who are unable to wear continuous monitoring due to a pacemaker or allergy.
* Patients who are not proficient in the Danish language will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of acceptability of the concept of wCVSM among orthopedic surgical ward nurses. | At 1, 6 and 12 months after post-implementation
  USE questionnaires will be distributed to the nurses taking care of patients undergoing ASD surgery.

SECONDARY OUTCOMES:
Assessment of acceptability of the concept of wCVSM in patients undergoing ASD surgery. | up to 7 days
  Patient acceptability will be measured cross-sectional by the System Usability Scale (SUS) questionnaire. SUS questionnaires will be distributed to the patients before discharge
Tecnical fidelity of the functioning of the continuous monitoring system | Up to 7 days
  Quantify total monitoring time, false positive alerts, false negative alerts and responses to alerts
Frequency of deviations in vital signs in patients after ASD surgery using wCVSM compared to NEWS2 | Up to 7 days
  The mean deviations detected per patient per day with wCVSM compared to deviations detected per patient per day with routine measurement.
Assessment of clinical outcomes after ASD surgery | Up to 30 days
  The mean surgical complications after ASD surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Joint surgery, University hospital, Rigshospitalet, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following publication of the manuscript and for five years afterwards
Access Criteria: Following publication of the manuscript, deidentified individual participant data will be available upon reasonable request. The project team will review each request on a case-by-case basis for a period of five years.